CLINICAL TRIAL: NCT00146445
Title: Intervention for Seropositive Injection Drug Users - Research and Evaluation (INSPIRE)
Brief Title: Behavioral Intervention Trial for HIV-infected Injection Drug Users
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Health Services Resource Adminstration - HIV/AIDS Bureau (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-2864; U22/CCU217990; U22/CCU317999; U22/CCU417998; U22/CCU918003
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: HIV
Keywords: IV drug users

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Peer Mentoring Intervention

SUMMARY:
The purpose of this study is to test whether a ten-session behavioral intervention for HIV-infected injection drug users is effective in reducing sex and injection risk behaviors that put others at risk for HIV infection, increasing access to or utilization of HIV primary health care, and increasing adherence to HIV medications.

DETAILED DESCRIPTION:
INSPIRE is a four-site (Baltimore, Miami, New York and San Francisco) randomized control trial to develop and evaluate the efficacy of a ten-session intervention for HIV-positive injection drug users. The primary goals of the intervention are to:

1. decrease sex and injection risk behaviors that put others at risk for HIV infection,
2. increase access to or utilization of HIV primary health care, and
3. increase adherence to HIV medications.

The intervention arm consists of 7 group sessions, 2 individual sessions, and one community experience. The control arm consists of 8 group sessions, aiming at controlling for demand (1st session) and attention (8 group sessions). Behavioral assessments and blood draws (for viral load and CD4 testing) occur at baseline, 6, and 12 month follow-up; a 3 month assessment involves behavioral assessment only. 1161 participants took baseline. Of these, 966 were randomized into the study, and 840, 807, and 821 participants took 3, 6, and 12 month follow-up assessments, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* self-identify as a person who has injected drugs in the last 12 months
* self-identify as a person who has had sex with at least one opposite sex partner within the last 3 months
* self-identify as HIV-seropositive
* be confirmed as HIV seropositive through oral fluid (saliva) HIV testing
* live in the geographic region under study,
* agree to have their blood drawn for CD4 count and viral load testing
* be willing to provide basic contact information (for follow-up)
* be able to communicate in English
* not have participated in the full-pilot of this intervention and not have enrolled previously in the present study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2001-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
- unprotected vaginal/anal sex with HIV-negative or unknown serostatus partners in the past 3 months
- lending needle or sharing cotton, cooker, or rinse water with HIV-negative or unknown serostatus partners in the past 3 months
-health care visits for HIV primary care in the past 6 months
-90% or more adherence to HIV medication yesterday and in the past week

SECONDARY OUTCOMES:
-Proportion of HIV status disclosure to sex partners

CONTACTS AND LOCATIONS:
Overall Officials: David W Purcell, JD, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (5):
- United States (5):
  - University of California - San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - New York Academy of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Background] Purcell DW, Metsch LR, Latka M, Santibanez S, Gomez CA, Eldred L, Latkin CA; INSPIRE Study Group. Interventions for seropositive injectors-research and evaluation: an integrated behavioral intervention with HIV-positive injection drug users to address medical care, adherence, and risk reduction. J Acquir Immune Defic Syndr. 2004 Oct 1;37 Suppl 2:S110-8. doi: 10.1097/01.qai.0000140609.44016.c4. PMID 15385907
- [Derived] Valverde EE, Purcell DW, Waldrop-Valverde D, Malow R, Knowlton AR, Gomez CA, Farrell N, Latka MH; INSPIRE Study Team. Correlates of depression among HIV-positive women and men who inject drugs. J Acquir Immune Defic Syndr. 2007 Nov 1;46 Suppl 2:S96-100. doi: 10.1097/QAI.0b013e318157683b. PMID 18089990
- [Derived] Mitchell SG, Edwards LV, Mackenzie S, Knowlton AR, Valverde EE, Arnsten JH, Santibanez S, Latka MH, Mizuno Y; INSPIRE Study Team. Participants' descriptions of social support within a multisite intervention for HIV-seropositive injection drug users (INSPIRE). J Acquir Immune Defic Syndr. 2007 Nov 1;46 Suppl 2:S55-63. doi: 10.1097/QAI.0b013e3181576808. PMID 18089985
- [Derived] Purcell DW, Latka MH, Metsch LR, Latkin CA, Gomez CA, Mizuno Y, Arnsten JH, Wilkinson JD, Knight KR, Knowlton AR, Santibanez S, Tobin KE, Rose CD, Valverde EE, Gourevitch MN, Eldred L, Borkowf CB; INSPIRE Study Team. Results from a randomized controlled trial of a peer-mentoring intervention to reduce HIV transmission and increase access to care and adherence to HIV medications among HIV-seropositive injection drug users. J Acquir Immune Defic Syndr. 2007 Nov 1;46 Suppl 2:S35-47. doi: 10.1097/QAI.0b013e31815767c4. PMID 18089983